CLINICAL TRIAL: NCT00066885
Title: A Phase 1/2 Multicenter, Open Label, Dose Ranging Study of DN-101 and Taxotere® in Patients With Advanced (Stage IIIB or IV) Non-Small Cell Lung Cancer (NSCLC) Who Have Failed Previous Therapy With Platinum-Based Chemotherapy
Brief Title: Study of DN101 and Taxotere in Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novacea (Industry)
Collaborators: Aventis Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DN101-004
Record Dates: First submitted 2003-08-06; First posted 2003-08-08 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2007-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: DN101; Calcitriol; Lung Cancer; NSCLC; Taxotere
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Calcitriol; Docetaxel

INTERVENTIONS:
Drug: calcitriol + docetaxel

SUMMARY:
This Phase 1/2 clinical trial is a multi-center, open-label study with three main objectives. The first (Phase 1A) is to determine the maximum-tolerated dose of DN-101 when administered in combination with Taxotere (docetaxel) every three weeks (closed). The second is to determine the maximum-tolerated dose of DN-101 when administered weekly in combination with Taxotere(docetaxel)devery three weeks (open). The third is to evaluate the safety and objective tumor response rate of the combination in NSCLC. DN-101 doses will be escalated at three dosing levels. Patients will receive oral DN-101 on day one, followed by intravenous docetaxel on day two of a 21-day cycle. Treatment cycles will be repeated at the same dose level each 21 days until disease progression or unacceptable toxicity.

DETAILED DESCRIPTION:
DN-101 is an oral anti-cancer therapy for solid tumors and various hematologic malignancies. DN-101 is a unique formulation of calcitriol specifically designed for use in cancer. Calcitriol is a naturally occurring hormone and the most potent biologically active form of vitamin D. In high doses, calcitriol is active in many laboratory and animal models of cancer and synergistic with many commonly used chemotherapeutic agents. Until recently, the clinical use of calcitriol as an anti-cancer therapy was limited by hypercalcemia at doses required for anti-tumor activity. Based upon clinical results to date, Novacea believes it has successfully developed a solution to this problem through development of DN-101.

Chemotherapy for NSCLC, while not curative, has been shown to prolong survival in patients with unresectable disease. A number of different chemotherapy agents have been shown to have single-agent activity in NSCLC. These include cisplatin, carboplatin, vinorelbine, gemcitabine, paclitaxel and docetaxel. For first-line therapy of Stage IIIB or Stage IV NSCLC, these agents are generally used in combination. In most cases, first-line chemotherapy consists of a platinum-based agent, either cisplatin or carboplatin, and another chemotherapeutic.

Only one agent, Taxotere®, has been approved in the United States by the Food and Drug Administration for use as second-line chemotherapy in NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically or cytologically proven non-small cell carcinoma of the lung (NSCLC), either Stage IIIB or Stage IV, that has progressed on or after first or second-line chemotherapy
* Measurable disease by RECIST criteria
* Eastern Cooperative Oncology Group (ECOG) Performance Status < 1
* Life expectancy > 3 months
* Age > 18 years
* Agrees to use adequate contraception throughout the treatment period and for at least 6 months following treatment
* Able to give informed patient consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2003-06; Study Completion 2005-12

CONTACTS AND LOCATIONS:
Overall Officials: Howard West, M.D., Study Chair — Swedish Cancer Institute
Locations (11):
- United States (11):
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - Kaiser Permanente Medical Center (Northern California), Vallejo, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - New York Oncology Hematology, P.C. - Albany Regional Cancer Center, Albany, New York
  - Piedmont Hematology Oncology Associates, PLLC, Winston-Salem, North Carolina
  - Cancer Care Associates, Tulsa, Oklahoma
  - Kaiser Permanente Northwest, Portland, Oregon
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Swedish Cancer Institute, Seattle, Washington
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
  - Yakima Regional Cancer Care Center, Yakima, Washington

REFERENCES:
- [Background] Beer TM, Eilers KM, Garzotto M, Egorin MJ, Lowe BA, Henner WD. Weekly high-dose calcitriol and docetaxel in metastatic androgen-independent prostate cancer. J Clin Oncol. 2003 Jan 1;21(1):123-8. doi: 10.1200/jco.2003.05.117. PMID 12506180